CLINICAL TRIAL: NCT02384720
Title: Study of Freefol-MCT PKPD in Healthy Volunteers
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Daewon Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: Freefol_PKPD_2013
Record Dates: First submitted 2015-02-24; First posted 2015-03-10 (Estimated); Last update posted 2016-10-10 (Estimated); Status verified 2016-10

CONDITIONS: Healthy
MeSH Terms: interventions — Aging

STUDY DESIGN:
Observational Model: Case-Only

GROUPS / COHORTS (3):
- A: Gender: 10 Males, 10 Females
  Interventions: Other: Age: 20-40years
- B: Gender: 10 Males, 10 Females
  Interventions: Other: Age: 41-64years
- C: Gender: 10 Males, 10 Females
  Interventions: Other: Age: ≥65years

INTERVENTIONS:
Other: Age: 20-40years
  Groups: A
Other: Age: 41-64years
  Groups: B
Other: Age: ≥65years
  Groups: C

SUMMARY:
The purpose of this study is to analysis PKPD of Freefol-MCT and to investigate relationship between the concentration of Freefol-MCT and the index which signaly analyzes those: EEG, EEG approximate entropy, systolic BP, saturation wave form and invasive BP wave form.

ELIGIBILITY:
Inclusion Criteria:

* Adults males/Females aged over 20years
* Health screening examination within 60 days of the start (Interview, vital signs , 12-lead ECG, blood tests, urinalysis) .
* The applicant who agreed in writing by told an explanation enough about the characteristics of the study drug, the purpose of the test and the details.

Exclusion Criteria:

* Subjects with clinically significant disease or history such as Liver, kidney, gastrointestinal, respiratory, musculoskeletal, endocrine, nervous psychiatric, blood tumor system and cardiovascular. (In particular, bronchial asthma, severe hepatic, renal failure, severe blood disorders, severe myasthenia gravis, cardiac dysfunction, peptic ulcer, etc.)
* Who had acute disease or organ dysfunction within four weeks of the start of the test.
* Who had significant hematologic disorders or donate whole blood within two months of the start of the test.
* Significant neuropsychiatric or more.
* Continued drug abuse.
* Who has a history of drug and other hypersensitivity reactions.
* Positive at Type B / C hepatitis , syphilis tests (VDRL), if in AIDS antibody test
* Who took other clinical medicine within two months of the start of the test.
* Who smokes or drinks within two weeks after dosing.
* Who takes drugs regularly other than the mineral claim or vitamin. However, it depends on judgment of the researchers.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy Adults over 20years old
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Primary Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Non- compartment pharmacokinetic parameters | 1200 minutes
Compartment pharmacokinetic parameters | 1200 minutes
BIS | 1200 minutes
SBP | 1200 minutes
E0 | 1200 minutes
Emax | 1200 minutes
Ce50 | 1200 minutes
ke0 | 1200 minutes